CLINICAL TRIAL: NCT04328129
Title: Household Transmission Investigation Study for Coronavirus Disease 2019 (COVID-19) in Tropical Regions
Brief Title: Household Transmission Investigation Study for COVID-19 in Tropical Regions
Acronym: EPI-COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut Pasteur de la Guyane (Unknown); Centre Hospitalier Andrée Rosemon de Cayenne (Unknown); Institut Pasteur de la Guadeloupe (Unknown); Centre Hospitalier de la Guadeloupe (Unknown); Institut Pasteur de Nouvelle-Calédonie (Unknown); Centre Hospitalier Territorial de Nouvelle-Calédonie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2020-009
Record Dates: First submitted 2020-03-23; First posted 2020-03-31 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Coronavirus Infections; Severe Acute Respiratory Syndrome; SARS-CoV Infection
Keywords: SARS-CoV-2; COVID-19; Serology; French Guiana
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary case (Experimental): Subject with laboratory-confirmed coronavirus SARS-CoV-2 infection by polymerase chain reaction (PCR)
  Interventions: Procedure: Human biological samples
- Family contact (Experimental): Subject who lived in the household of the primary case while the primary case was symptomatic
  Interventions: Procedure: Human biological samples

INTERVENTIONS:
Procedure: Human biological samples — * Blood sample
  * Nasopharyngeal swab.

SUMMARY:
This study is a interventional study that present minimal risks and constraints to evaluate the presence of novel coronavirus (SARS-CoV-2) or antibodies among individuals living in households where there is a confirmed coronavirus case in order to provide useful information on the proportion of symptomatic forms and the extent of the virus transmission in tropical regions such as French Guiana, Guadeloupe and New-Caledonia.

DETAILED DESCRIPTION:
This study is a interventional study that present minimal risks and constraints to evaluate the presence of novel coronavirus (SARS-CoV-2) or antibodies among individuals living in households where there is a confirmed coronavirus case in order to provide useful information on the proportion of symptomatic forms and the extent of the virus transmission in tropical regions such as French Guiana, Guadeloupe and New-Caledonia.

Subjects will be assessed (questionnaires and sampling) in their homes. Subjects will be asked to attend study visits at days 0, 7, 14, 21, 28, 60, 90, 180 and 360.

The primary objective of the study is to evaluate the rate of intra-household secondary transmission of the virus.

ELIGIBILITY:
Inclusion Criteria:

* Primary case: laboratory-confirmed coronavirus SARS-CoV-2 infection by polymerase chain reaction (PCR),

or Family contact in French Guiana and Guadeloupe: person who lived in the same household as the primary case of COVID-19 when the primary case was symptomatic. A household is defined as a group of people (2 or more) living in the same accommodation (excluding residential institutions such as boarding schools, dormitories, hostels, prisons, other communities hosting grouped people),

or Close contact in New-Caledonia: any individual who was in contact with a primary case, in his/her family/living environment, work/school, friends/leisure or means of transport, when the primary case was symptomatic or presymptomatic,

* Affiliated or beneficiary of a social security system
* Informed consent prior to initiation of any study procedures from subject (or legally authorized representative)
* State of health compatible with a blood sample as defined in the protocol.

Exclusion Criteria:

* Inability to consent
* Person under guardianship or curatorship
* Known pathology or a health problem contraindicated with the collect of blood sample.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the extent of the virus transmission within households | 2 years
  The extent of the virus transmission within households will be assessed by evaluating the rate of intra-household secondary transmission of the virus

SECONDARY OUTCOMES:
Characterization of the secondary cases | 2 years
  The characterization of the secondary cases will be assessed by evaluating the proportion of asymptomatic forms within the household
Characterization of the secondary cases | 2 years
  The characterization of the secondary cases will be assessed by characterizing the risk factors for coronavirus infection.
In New-Caledonia, evaluation of the extent of the virus transmission within contact persons | 2 years
  The extent of the virus transmission within contact persons will be assessed by evaluating the rate of extended-contact secondary transmission of the virus

CONTACTS AND LOCATIONS:
Overall Officials: Claude Flamand, PhD, Principal Investigator — Institut Pasteur de la Guyane, Head of Epidemiology Unit
Locations (4):
- French Guiana (2):
  - Centre Hospitalier Andrée Rosemon, Cayenne
  - Institut Pasteur de la Guyane, Cayenne
- Institut Pasteur de Guadeloupe, Les Abymes, Guadeloupe
- Institut Pasteur de Nouvelle-Calédonie, Noumea, New Caledonia

IPD SHARING:
Plan to Share IPD: No